CLINICAL TRIAL: NCT02217735
Title: Randomized Controlled Expressive Writing Pilot in Individuals With Parkinson's Disease and Their Caregivers
Brief Title: Expressive Writing for Individuals With Parkinson's Disease and Their Caregivers
Acronym: PDEWS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM#13659
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Parkinson's Disease; Coping Skills
Keywords: Parkinson's Disease; Caregivers; Expressive Writing; Complementary Medicine; Cortisol
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Writing Intervention - Expressive Arm (Experimental): Participants are asked to write about the most traumatic or stressful experience of their entire lives in three, 20 minute writing sessions.
  Interventions: Behavioral: Writing Intervention
- Writing Intervention - Neutral Arm (Active Comparator): Participants are asked to write about what they did the day before, refraining from including emotional details.
  Interventions: Behavioral: Writing Intervention

INTERVENTIONS:
Behavioral: Writing Intervention — Participants wrote for 20 minutes on three occasions about an emotional or traumatic topic (expressive writing intervention condition) or what they did the day before, while refraining from including emotional details.

SUMMARY:
This randomized, controlled trial (RCT) evaluates the benefits of expressive compared to neutral writing in individuals with Parkinson's Disease and their support persons. Participants will be randomly assigned to complete three, 20 minute sessions of expressive or neutral writing. Participants will complete evaluation of outcomes at baseline, immediate post, 4 month and 10 month follow ups to establish if benefits remain over time. Impact of these therapies on thinking abilities, physical health, and patient and support person ratings of thinking skills, mood and quality of life will be evaluated. Expressive writing is hypothesized to result in greater improvements and/or stability of function on neuropsychological tests of attention, working memory, learning, and memory skills compared to the neutral writing condition.

Results from this study will determine whether brief writing exercises are easily used by and beneficial for individuals with Parkinson's Disease and their support persons. If positive benefit is observed, information from this study will be used to further optimize these therapies for larger trials designed to evaluate the value of the therapies for individuals with Parkinson's Disease and their support persons.

DETAILED DESCRIPTION:
The expressive writing condition asks participants to write about the most stressful or traumatic experience of their entire lives over three, 20 minute private writing sessions. The neutral control writing conditions asks participants to write about how they spent their time the day before.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Parkinson's Disease Caregiver of an individual with Parkinson's Disease

Exclusion Criteria:

Clinical diagnosis of Dementia Clinical diagnosis of other Parkinson's Disease-associated comorbid conditions (e.g., severe anxiety, depression, excessive daytime sleepiness, or psychosis) that significantly influence cognitive testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Quality of Life (PDQ-39) | Baseline to immediate post

SECONDARY OUTCOMES:
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | Immediate post to 4-month follow up
Parkinson's Disease Quality of Life Questionnaire (PDQ-39) | 4 month follow up to 10 month follow up

OTHER OUTCOMES:
Expressive Writing | three samples collected during the intervention period (which occurs between baseline and immediate post assessments)
  The three writing samples from each participant in the Expressive Arm will be qualitatively examined for themes about traumatic events.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K. Lageman, Ph.D., Principal Investigator — Virginia Commonwealth University; James P. Bennett, M.D., Ph.D., Study Chair — Virginia Commonwealth University
Locations (1):
- VCU Parkinson's and Movement Disorders Center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Cash TV, Lageman SK. Randomized controlled expressive writing pilot in individuals with Parkinson's disease and their caregivers. BMC Psychol. 2015 Nov 30;3:44. doi: 10.1186/s40359-015-0101-4. PMID 26621025